CLINICAL TRIAL: NCT02797275
Title: Lung Anatomic, Physiologic, and Inflammatory Changes With Chronic Exposure to Secondhand Tobacco Smoke
Brief Title: Secondhand Smoke Respiratory Health Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Flight Attendant Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SHS; 13631 (Other: University of California, San Francisco)
Record Dates: First submitted 2016-05-06; First posted 2016-06-13 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Secondhand Smoke; Air Trapping; Tobacco; Airflow Limitation; Hyperinflation; Obstructive Lung Disease
MeSH Terms: conditions — Lung Diseases, Obstructive | interventions — Albuterol; Procaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albuterol & Placebo (Experimental): Participants will be placed on the albuterol treatment (2 puffs twice a day, equivalent to 360 mcg per day) after the completion of the baseline screening visit. They will use albuterol for 4 weeks prior to their scheduled second visit during which they will undergo testing. Subsequently, and after a minimum washout period of 2 weeks, they will be placed on the placebo treatment for 4 weeks prior to their scheduled third visit, after which they will come back to undergo testing.
  Interventions: Drug: Albuterol; Drug: Placebo
- Placebo & Albuterol (Experimental): Participants will be placed on the placebo treatment after the completion of the baseline screening visit. They will use placebo for 4 weeks prior to their scheduled second visit during which they will undergo testing. Subsequently, and after a minimum washout period of 2 weeks, they will be placed on the albuterol treatment (2 puffs twice a day, equivalent to 360 mcg per day) for 4 weeks prior to their scheduled third visit, after which they will come back to undergo testing.
  Interventions: Drug: Albuterol; Drug: Placebo

INTERVENTIONS:
Drug: Albuterol — Beta agonist respiratory inhaler
  Other Names: ProAir
Drug: Placebo — respiratory inhaler with no medication
  Other Names: Placebo obtained from Teva

SUMMARY:
Exposure to secondhand tobacco smoke (SHS) is associated with diverse health effects in nonsmokers. Flight attendants (FA) who worked on commercial aircraft before the ban on tobacco smoking (exposed FAs) had high, long-term levels of occupational exposure to SHS and are a unique population for the study of long-term health effects of chronic exposure to SHS.

In previous studies, we have shown that many never-smoking SHS-exposed FAs to have curvilinear flow-volume loops, decreased airflow at mid- and low-lung volumes, and static air trapping (elevated residual volume to total lung capacity ratio [RV/TLC]), abnormalities that are not diagnostic of overt Chronic Obstructive Pulmonary Disease (COPD), but do implicate the presence of an obstructive ventilatory defect, and are consistent with what has been recently described as preserved ratio impaired spirometry (PRISm).

The main objective of the study is to determine the effect of a bronchodilator to counter the physiologic abnormalities that are observed in the population of never-smoking SHS-exposed FAs as both proof of concept of the presence of an obstructive lung disease and as a possible therapeutic option to counteract the adverse respiratory effects of chronic exposure to SHS.

DETAILED DESCRIPTION:
The objective of this research plan is to investigate the hypothesis that subclinical airflow limitation and air trapping in never-smoking SHS-exposed individuals with preserved ratio impaired spirometry (PRISm) causes reduced exercise capacity . This in turn will adversely affect their symptoms and quality of life. Furthermore, we hypothesize that exercise capacity, symptoms, and quality of life will improve with the use of inhaled bronchodilators.

We proposed to investigate the above hypotheses through the following specific aims:

Aim 1- Determine whether airflow limitation in never-smoking SHS-exposed individuals with airflow limitation or air trapping is associated with reduced exercise capacity and adverse health and health-related quality of life (HRQL). We propose to measure (1) maximum level of exercise (watts) and maximum oxygen uptake (VO2) in the laboratory setting, (2) level of physical activity during the subjects' routine daily life using an activity monitor, and (3) measure HRQL using survey tools. We propose to then explore associations between these measures and indices of air trapping at rest (RV/TLC) and progressive airflow limitation with exercise (end expiratory lung volume (EELV)and dynamic hyperinflation (DH)).

Aim 2: Determine whether relief of airflow limitation using bronchodilators could improve exercise capacity in never-smoking SHS-exposed individuals with airflow limitation or air trapping in a double blind crossover placebo-controlled randomized clinical trial. We propose to examine the effect of bronchodilators on airflow limitation and air trapping and their effects in turn on exercise capacity, daily level of physical activity, and HRQL to show a cause-and-effect relationship. In this way, we plan to explore the utility of bronchodilators as a treatment option for the observed reduced exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Never Smoking SHS-exposed Flight Attendants:

   * aircraft cabin SHS exposure of >1 year while working for airlines
   * Never smoker as defined by use of <100 cigarettes lifetime and none within the last year.
   * Normal forced expiratory volume (FEV) FEV1/ forced vital capacity (FVC) ratio
   * One of the following evidence of airflow obstruction:

     * Presence of any airflow limitation on spirometry during the baseline visit
     * Development of airflow limitation on spirometry during any stages of exercise testing
     * Residual volume to total lung capacity ratio of >0.35
2. Exclusion Criteria:

   * History of active cardiac disease, uncontrolled hypertension, congestive heart failure
   * History of direct tobacco use of over 100 cigarettes in their lifetime
   * History of established respiratory diseases such as asthma, emphysema, chronic bronchitis, interstitial lung disease, or sarcoidosis
   * History of debilitating chronic illnesses such as severe lupus or rheumatoid arthritis
   * History of other illnesses or therapy for illnesses that could affect lung function such as radiation therapy for breast cancer
   * Physical inability to perform exercise testing
   * BMI >30 kg/m2
   * History of marijuana use of >100 joints lifetime, and none within the last year
   * History of other recreational drug use

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Oxygen Consumption (Max VO2) | 4 weeks
  Maximum oxygen consumption (Max VO2) as determined by a symptom-limited progressively increasing cycle exercise test to determine the maximum work (watts) and oxygen uptake (VO2) achieved. The protocol consisted of 3-min rest, 1-min unloaded (freewheeling) cycling at 60 rpm, followed by increasing work rate of 20-30 Watts each 2 minutes to a maximum tolerated, and 5-min of recovery. Twelve lead ECGs were monitored continuously and were recorded along with BP every 2 min. Oxyhemoglobin saturation (O2sat) determined by pulse oximetry was recorded continuously.

SECONDARY OUTCOMES:
Airflow Limitation | 4 weeks
  After 30 minutes period of rest, the subject will perform exercise at increasing work rates corresponding to 20%, 40%, 60%, and 80% of the maximum oxygen uptake attained in the first exercise with 2 minutes at each stage. Inspiratory capacity will be measured 2 to 3 times at each work rate while recording tidal flow-volume loops to assess for evidence of airflow limitation during exercise. Air flow limitation will be determined by calculating the percent overlap of tidal breathing over expiratory portion of maximum flow.
Dynamic Hyperinflation | 4 weeks
  After 30 minutes period of rest, the subject will perform exercise at increasing work rates corresponding to 20%, 40%, 60%, and 80% of the maximum oxygen uptake attained in the first exercise with 2 minutes at each stage. Inspiratory capacity will be measured 2 to 3 times at each work rate while recording tidal flow-volume loops to assess for evidence of airflow limitation during exercise. Dynamic hyperinflation will be measured by changes in examining end-expiratory lung volume at each stage.
Change in scores on the SF-12® Health Survey Short Form (SF-12) | Up to 12 months
  The SF-12 is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective. The SF-12 consists of a subset of 12 items from the SF-36® Health Survey (SF-36) and measures two composite outcomes assessing mental health composite score (MCS) and physical health composite scores (PCS). The PCS & MCS are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The absolute change in item score by group from baseline up to 12 months was used to assess the quality of life/psychosocial impact on the patients with a larger scores indicating a greater degree of change on physical and mental health.
Change in scores on the Airway questionnaire (AQ20) | Up to 12 months
  The AQ20 is given to patients to measure HRQOL related to asthma and chronic obstructive pulmonary disease (COPD) . It contains 20 items, with scores ranging from 0 to 20 - high scores indicate poor HRQOL. The absolute change in item score by group from baseline up to 12 months will be reported
Change in scores on the International Physical Activity Questionnaires (IPAQ) | Up to 12 months
  The IPAQ measure a participants physical activity by either telephone interview or self-administered methods. IPAQ assesses physical activity undertaken across a comprehensive set of domains including: leisure time physical activity, domestic and gardening (yard) activities, work-related physical activity, and transport-related physical activity. Based on the participant responses, results are categorized into Low, Moderate, or High levels of physical activity. The absolute change in score by group from baseline up to 12 months will be reported
Change in level of physical activity over time | Up to 12 months
  Real world (outside lab) level of physical activity will be measured using an activity monitor (Actigraph) over a period of a week starting the third week during their treatment. The Actigraph is a monitor that allows collection and analysis of daily activity information about subjects in their normal daily living environment, which records both the number of steps and the time interval during which the steps are taken. The change in score by group from baseline up to 12 months will be reported
Association between respiratory abnormalities and HRQOL outcomes. | Up to 12 months
  The association between respiratory abnormalities and HRQOL outcomes at 12 months will be determined using pearson/spearman correlation. The aim is to show that at least 8%-10% of the variation in level of physical activity or score on our survey tools are explained by the observed lung function abnormalities and cabin SHS exposure (a correlation coefficient of at least 0.28). Correlation coefficients range from + 1 to -1, with a coefficient of 0=no correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Arjomandi, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - VA Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT02797275/ICF_000.pdf